CLINICAL TRIAL: NCT05207540
Title: A Reliability and Validity Study of Urdu Version Of Cornell Musculoskeletal Discomfort Questionnaire
Brief Title: Urdu Version Of Cornell Musculoskeletal Discomfort Questionnaire: Reliability And Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00299
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Musculoskeletal Pain
Keywords: Cornell musculoskeletal discomfort questionnaire; factory workers; reliability; validity; Musculoskeletal discomfort
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to translate and adapt Cornell Musculoskeletal Discomfort Questionnaire cross-culturally into the Urdu language for the Pakistani population for investigating the reliability and validity of Cornell Musculoskeletal Discomfort Questionnaire in the Pakistani population and to study the correlation between Nordic Musculoskeletal Questionnaire and the Visual Analogue Scale.

DETAILED DESCRIPTION:
The English version of the Cornell Musculoskeletal Discomfort Questionnaire will be translated into Urdu and culturally adapted, as per a previous recommendation. The Cornell Musculoskeletal Discomfort Questionnaire will be given to one hundred and fifty workers of Masood Textile Mills, who would be chosen based on convenience sampling and inclusion and exclusion criteria. The inter-observer and intra-observer reliability of the Cornell Musculoskeletal Discomfort Questionnaire, Nordic Musculoskeletal Questionnaire, and Visual Analog Scale will be evaluated in this study. On the same day, the questionnaire will be filled out created two times. An Inter - observer assessment will be done with 2 hour break between distributions of questionnaires. The initial observer then will gather a third assessment over one-week period (intra-observer assessment). For data entry and analysis, Statistical Package of Social Sciences Version 24 will be utilized. Internal consistency will be checked using the Cronbach alpha value, and test retest reliability will be assessed using the Intraclass coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Participants having an age limit of 18 to 55.
* Could read and understand the Urdu language.
* Both males and females working more than 6 hours in sitting and standing positions.

Exclusion Criteria:

* Having any fracture in any part of the body.
* Having any congenital or acquired disability that restricts them in their daily living.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population suffering from musculoskeletal discomfort with a working routine of more than 6 hours both in sitting and standing position.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal Discomfort Questionnaire | 1st day
  This questionnaire is used to access discomfort caused by Musculoskeletal disorders. It has 3 scales, frequency, severity and interference scale. It has 3 versions on the basis of the nature of work place and activity level i.e. Sedentary workers, standing workers and hand discomfort. Sedentary workers don't include the "foot" domain while the standing worker has this domain. The hand discomfort version is used to access only hand problems. Its interpretation can be done by multiplying all the scale score.
Nordic Musculoskeletal Questionnaire | 1st day
  The Nordic Questionnaire is an internationally recognized tool for standardization research on Musculoskeletal symptom assessment. Its goal is to use an ergonomically approach to analyze Musculoskeletal problems. The very first component of this instrument includes questions on body parts that correlate to nine anatomical regions. The questions were structured in the following sequence: yearly and weekly prevalence; functional disability; and seeking medical treatment in the last year. This questionnaire can be used in an examination or by the individual who is now being assessed.
Visual Analogue Scale | 1st day
  The Visual Analogue Scale was created to represent the concept of a fundamental continuity. A Visual Analogue Scale is typically a straight stripe measuring 100 mm long, with word descriptions for each end. The patient draws a line through the spot on the line which they believe best describes their present state. The Visual Analogue Scale score is calculated by calculating in millimeters as from the line's left side to the point marked by that of the patient. It usually ranges from "0" indicating "no pain" to the "10" indicating "worst pain".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No